CLINICAL TRIAL: NCT07205523
Title: High-Altitude Hematology Observation-Stem Cell Transplantation (HALO-SCT): A Prospective Real-World Cohort Study in the Qinghai-Tibet Plateau
Brief Title: High-Altitude Hematology Observation-Stem Cell Transplantation (HALO-SCT)
Acronym: HALO-SCT
Status: Recruiting | Type: Observational
Sponsor: Yigeng Cao,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Yigeng Cao,MD,PhD, Affiliated Hospital of Qinghai University, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Other Study IDs: HALO-SCT-2023
Record Dates: First submitted 2025-09-12; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic Stem Cell Transplantation (HSCT); Acute Myeloid Leukemia (AML); Leukemias, Acute Myeloid; Myeloid Leukemias, Acute; Hemophilia; Myelodysplastic Syndrome; MDS; Lymphoma; Leukemia; Aplastic Anemia; Bleeding Disorders; Bone Marrow Transplantation; Multiple Myeloma; Myeloma, Multiple; Immune Reconstitution
Keywords: High-altitude Bone marrow transplantation Allogeneic HSCT Autologous HSCT Immune reconstitution Graft-versus-host disease Relapse Survival Quality of life
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hemophilia A; Myelodysplastic Syndromes; Lymphoma; Leukemia; Anemia, Aplastic; Hemostatic Disorders; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSCT Patients and Donors: Patients undergoing hematopoietic stem cell transplantation (HSCT) at Qinghai University Affiliated Hospital, and their related or unrelated stem cell donors. Participants are prospectively followed for clinical outcomes and biospecimen collection under real-world conditions.

SUMMARY:
The High-Altitude Hematology Observation-Stem Cell Transplantation (HALO-SCT) study is the first prospective real-world cohort of hematologic diseases and transplantation in the Qinghai-Tibet Plateau. Patients undergoing hematopoietic stem cell transplantation (HSCT) at Qinghai University Affiliated Hospital, together with their donors, are systematically enrolled. The registry collects demographic, diagnostic, treatment, prognosis, and medical expense information, as well as biospecimens for future analyses. Historical data are incorporated, and prospective data collection is ongoing with long-term follow-up planned. The registry is designed as a sustainable research infrastructure to provide comprehensive data on disease incidence, treatment patterns, outcomes, and resource utilization in a high-altitude setting.

DETAILED DESCRIPTION:
HALO-SCT is a prospective observational patient registry established at Qinghai University Affiliated Hospital, the first HSCT center in the Qinghai-Tibet Plateau. The registry aims to systematically capture patient and donor characteristics, transplant-related procedures, treatment outcomes, and long-term follow-up data in a high-altitude environment. Biospecimens, including peripheral blood and bone marrow samples, are collected at baseline and follow-up time points for future multi-omics studies. All clinical decisions follow routine practice; no experimental interventions are mandated by the protocol. The registry is intended as a long-term infrastructure project, with continuous data collection and integration into national and international collaborative research efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with hematologic diseases who are admitted to the HSCT center of Qinghai University Affiliated Hospital on or after September 1, 2023.
2. Planned or actual hematopoietic stem cell transplantation (HSCT).
3. Provision of signed informed consent.

Exclusion Criteria:

1. Inability to provide long-term follow-up data due to severe comorbidities or logistical reasons.
2. Substance abuse compromising adherence.
3. Any condition judged by investigators to jeopardize safety or compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematologic diseases undergoing hematopoietic stem cell transplantation (HSCT) and their donors at the Affiliated Hospital of Qinghai University, located in the Qinghai-Tibet Plateau. The registry systematically captures demographic, clinical, and outcome data under real-world conditions in a high-altitude environment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2060-12-31 (Estimated); Study Completion 2100-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | From the date of HSCT until neutrophil engraftment or death, assessed up to 60 days
  Defined as the first of 3 consecutive days with absolute neutrophil count (ANC) ≥ 0.5 × 10⁹/L without primary graft failure. Patients who die without engraftment before day +60 will be censored.

SECONDARY OUTCOMES:
Incidence of acute GVHD | From the date of HSCT until day +100, assessed up to 100 days
  Proportion of patients developing grade I-IV acute GVHD, excluding events occurring after donor lymphocyte infusion (DLI). Diagnosis and grading based on consensus criteria (e.g., MAGIC).
Overall survival | From the date of HSCT until death from any cause, assessed up to 12 months
  OS is defined as time from HSCT to death from any cause. Patients alive at last follow-up will be censored.
Disease-free survival | From the date of HSCT until relapse/progression or death from any cause, whichever occurs first, assessed up to 12 months
  DFS is defined as survival without relapse or progression. Patients alive without relapse at last follow-up will be censored.
Cumulative incidence of relapse | From the date of HSCT until relapse/progression, assessed up to 12 months
  Cumulative incidence of relapse/progression, with non-relapse mortality treated as a competing risk.
Immune reconstitution | From the date of HSCT until 12 months post-transplant, assessed at prespecified time points (e.g., day +30, +180,)
  Serial assessment of immune reconstitution, including lymphocyte subsets, immunoglobulin recovery, and functional immune assays.
Incidence of chronic GVHD | From the date of HSCT until 12 months post-transplant, assessed up to 12 months
  Proportion of patients developing chronic GVHD, diagnosed and graded according to NIH 2014 consensus criteria. Death and relapse treated as competing risks.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Geng, Principal Investigator — Affiliated Hospital of Qinghai University
Locations (1):
- Affiliated Hospital of Qinghai University, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the registry collects sensitive clinical and genetic information from transplant patients and donors in a high-altitude region. Data sharing may compromise patient privacy and is not permitted under current institutional and ethical committee policies. Only aggregated results will be reported publicly.